CLINICAL TRIAL: NCT06244758
Title: Effects of Finerenone on Renal Hemodynamics and Oxidative Stress
Brief Title: Finerenone and Renal Oxidative Stress
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FINE
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Type2diabetes
MeSH Terms: interventions — finerenone; Tablets

STUDY DESIGN:
Intervention Model Description: randomized (1:1), prospective, double-blind, placebo controlled, parallel-group, single centre study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): Renal hemodynamic parameters and oxidative stress will be obtained and the patient will be given finerenone orally
  Interventions: Drug: Finerenone 20 MG Oral Tablet
- Placebo (Placebo Comparator): Renal hemodynamic parameters and oxidative stress will be obtained and the patient will be given placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone 20 MG Oral Tablet — The intervention is administered orally.
  Arms: Treatment
Drug: Placebo — The intervention is administered orally.
  Arms: Placebo

SUMMARY:
The main goal of this mechanistic, prospective, double-blind, placebo controlled, randomized study is to demonstrate the effect of finerenone on the oxidative stress of renal vasculature. Moreover, parameters of renal hemodynamics like renal plasma flow, total renal vascular resistance, filtration fraction, parameters of intraglomerular hemodynamics etc. are analyzed in detail. Finally, the change in renal nitric oxide activity with finerenone treatment is analyzed.

The primary objective of this mechanistic study is to analyse:

- the impact of finerenone on the oxidative stress level of renal vasculature by the increase of renal perfusion following vitamin C infusion compared to placebo

DETAILED DESCRIPTION:
Non-traditional risk factors such as oxidative stress and inflammation are highly prevalent in patients with chronic kidney disease, cardiovascular disease and diabetes mellitus. Diabetes mellitus, which is considered at the beginning as a metabolic disorder, converts rapidly into a predominantly vascular disease. Hyperglycemia upregulates markers of chronic inflammation and contribute to increased reactive oxygen species generation, which ultimately cause vascular dysfunction. Endothelial dysfunction occurs early in the process of vascular impairment. One of the potential mechanisms contributing to endothelial dysfunction in diabetic patients is inactivation of nitric oxide by oxygen-derived free radicals. Similarly, oxidatively mediated degradation of endothelium-derived nitric oxide contributing to abnormal endothelium-dependent vasodilation has been observed in animal models of diabetes mellitus. Similar mechanisms are associated with early chronic kidney disease and its progression. Indeed, studies in animal models have demonstrated that administration of antioxidants restores normal endothelial function.

In patients with CKD and type 2 diabetes, treatment with finerenone resulted in lower risks of CKD progression and cardiovascular events than placebo (FIDELIO, FIGARO studies and FIDELITY analysis). Preclinical data showed that the kidney and cardiovascular benefits of finerenone were associated with potent anti-inflammatory and antifibrotic effects through inhibition of overactivation of the mineralocorticoid receptor. Blockade of the mineralocorticoid receptor with finerenone may reduce production of reactive oxygen species, observed to be increased in diabetes already at the early stage as well as in patients with overt nephropathy. However, there is no study in humans supporting this mechanism how finerenone may exert nephroprotective effects. This mechanistic study attempts to support this concept with in vivo data in patients.

Vitamin C is a water-soluble antioxidant capable of scavenging free radicals and was found to restore the impaired endothelium-dependent vasodilation in the forearm resistance vessels of patients with diabetes mellitus. The investigators previously examined the role of oxidative stress in the renal circulation in humans by measuring the response of Vitamin C on renal plasma flow with constant clearance input technique. The investigators observed first that vitamin C reduced the high level of oxidative stress in the renal vasculature in smokers known to have increased oxidative stress. Subsequently, the investigators found in patients with type 2 diabetes with normal renal function that the increase of renal plasma flow following vitamin C infusion is augmented in type 2 diabetes indicating increased formation of reactive oxygen species already in the early stage of diabetic disease. Finally, the investigators also found infusion of the antioxidant vitamin C (on top of L-arginine) induced a more pronounced increase in renal plasma flow in patients with chronic kidney disease than in control subjects. All these previous studies allowed us to conclude that vitamin C infusion is a tool to measure oxidative stress of the renal vasculature in humans in vivo, which clearly contrasts the measurement of biomarkers in the urine or peripheral blood samples. In addition, the infusion of L-arginine, a substrate for nitric oxide synthesis, emerged in our hands as a tool to measure nitric oxide synthesis in the renal circulation, since the vasodilatory response to L-arginine, at least in part, was due to increased production and release of nitric oxide. Thus, the bioavailability of nitric oxide can be judged by measuring the change of renal plasma flow to L-arginine infusion in addition to measure albuminuria.

Patients with type 2 diabetes are an ideal study population to analyze any effect of an intervention on oxidative stress and nitric oxide bioactivity since hyperglycemia upregulates markers of chronic inflammation and contributes to increased reactive oxygen species already in the prediabetes stage, far before renal function or cardiovascular atherosclerotic processes become clinically overt. Our data in patients with type 2 diabetes who had normal renal function support this notion. Effects of finerenone on oxidative stress are therefore measurable in this early stage of type 2 diabetes. Furthermore, our so far used model of measuring oxidative stress (by vitamin C infusion) and stimulated nitric oxide bioactivity (by L-arginine infusion) in the renal circulation has been validated for eGFR >45 ml/min/1.73m² and our findings were consistently found in type 2 diabetes as well as in patients with diagnosed chronic kidney disease.

The investigators use the constant input clearance technique, considered globally as gold standard to analyze renal function, with para-amino-hippuric acid (PAH) for the measurement of renal plasma flow and iohexol (inulin and sinestrin are no longer available) for the measurement of glomerular filtration rate. The investigators therefore avoid any inaccuracy related to incomplete urine sampling and complete bladder voiding. In addition, the investigators apply the Gomez formula to estimate intraglomerular pressure and afferent and efferent glomerular resistances. This is possible if the Gomez formula are applied to measurements in patients with only minor altered renal morphology (i.e normal renal function). To our knowledge, no detailed analysis of renal hemodynamics, including intraglomerular resistances, are available for finerenone in humans. A decrease of the intraglomerular pressure could be an additional explanation of the beneficial nephroprotective effects of finerenone. Please note that the investigators have used this technique as part of several studies and clinics (for example to analyze the exact renal function in potential kidney donors) since more than 20 years.

Infusion of L-arginine permits the assessment of stimulated nitric oxide dependent vasodilation in the renal circulation (and thereby of nitric oxide bioavailability) by measuring the change of renal plasma flow to L-arginine infusion. The dose of L-arginine at 100mg/kg (in contrast to 250 and 500 mg/kg) was found to be the most suitable dose, because of the absence of any systemic hemodynamic changes and the absence of direct osmotic effects of any amino acid load (in contrast to 500 mg/kg). Infusion of the antioxidant vitamin C (on top of L-arginine) allows us to reduce in vivo the level of oxidative stress, and the increase in RPF due to vitamin infusion is an estimate of the oxidative stress in the renal vasculature at baseline. For details see our previous work. So far, there are no clinical data or an in-depth analysis (in vivo) of the effects on renal hemodynamics after treatment with finerenone. In-Vivo data supporting the concept that finerenone improves renal hemodynamics, oxidative stress, renal nitric oxide activity is lacking, and our study aims at closing this knowledge gap by measuring various renal parameters following infusion of vitamin C and L-arginine thereby allowing us to delineate a complete profile of the renal effects of finerenone. Such an approach is now in particular of relevance since the European Medicines Agency (EMA) has already approved finerenone (Kerendia®) within the EU.

Our hypothesis is that in face of its impressive nephroprotective effect finerenone exerts beneficial effects on renal hemodynamics by reducing renal oxidative stress. The main goal of this mechanistic, prospective, double-blind, placebo controlled, randomized study is to demonstrate the effect of finerenone on the oxidative stress of renal vasculature. Moreover, parameters of renal hemodynamics like renal plasma flow, total renal vascular resistance, filtration fraction, parameters of intraglomerular hemodynamics etc. are analyzed in detail. Finally, the change in renal nitric oxide activity with finerenone treatment is analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 75 years
* Diagnosis of type 2 diabetes mellitus (defined by ADA criteria)
* Male and Female patients (females of child bearing potential must be using effective contraceptive precautions per CTFG quidance)
* Females of childbearing potential or within two years of the menopause must have a negative urine pregnancy test at screening visit
* Informed consent (§ 40 Abs. 1 Satz 3 Punkt 3 AMG) must be given in written form

Exclusion Criteria:

* Any other form of diabetes mellitus than type 2 diabetes mellitus
* Female who is pregnant, breast feeding or intends to become pregnant. Documentation of highly effective contraception is required for women of childbearing potential. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for 3 months after stopping medication
* Use of insulin or GLP-1 analogue within the past 3 months
* HbA1c ≥ 10.5%
* Serum potassium > 4.8 mmol/l
* Body mass index > 40 kg/m²
* Estimated glomerular filtration rate (eGFR) < 45 ml/min/1.73m² (CKD-EPI Formula)
* Uncontrolled arterial hypertension (BP ≥ 180/110 mmHg)
* Subclinical or clinical hyperthyroidism
* Significant laboratory abnormalities such as serum Glutamate-Oxaloacetate-Transaminase (SGOT) or serum Glutamate-Pyruvate-Transaminase (SGPT) levels more than 3 x above the upper limit of normal range
* Use of strong CYP3A4-Inhibitors (for example Itraconazol, Clarithromycin, Ketoconazol, Ritonavir, Nelfinavir, Cobicistat, Telithromycin, Nefazodon) or CYP3A4-Inducers (for example Rifampicin, Carbamazepin, Phenytoin, Phenobarbital, St. John's wort (Johanniskraut), Efavirenz)
* Use of other aldosterone receptor antagonist like spironolactone or eplerenone or potassium sparing diuretics or direct renin inhibitors
* Any history of stroke, transient ischemic attack, instable angina pectoris, or myocardial infarction within the last 6 months prior to study inclusion
* Congestive heart failure (CHF) NYHA stage IV
* Drug or alcohol abuse
* Severe disorders of the gastrointestinal tract or other diseases which interfere with the pharmacodynamics and pharmacokinetics of the study drug
* Allergic reaction to iodine
* Individuals at risk for poor protocol or medication compliance
* Participation in another clinical study within 30 days prior to visit 1
* Patients being treated for severe auto immune disease e.g. lupus, glomerulonephritis
* Any patient currently receiving chronic (>30 consecutive days) treatment with an oral corticosteroid - Patients in unstable conditions due to any kind of serious disease, that interferes with the conduct of the trial
* Subject who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 GCP-V

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the impact of finerenone on the oxidative stress level of renal vasculature by the increase of renal perfusion following vitamin C infusion compared to placebo | at baseline and after 3 months on finerenone
  the impact of finerenone on the oxidative stress level of renal vasculature by the increase of renal perfusion following vitamin C infusion compared to placebo

SECONDARY OUTCOMES:
impact of finerenone on renal plasma flow (para-aminohippurate (PAH) clearance) compared to placebo | at baseline and after 3 months on finerenone
  impact of finerenone on renal plasma flow (para-aminohippurate (PAH) clearance) compared to placebo
impact of finerenone on glomerular filtration rate (iohexol clearance) compared to placebo | at baseline and after 3 months on finerenone
  impact of finerenone on glomerular filtration rate (iohexol clearance) compared to placebo
impact of finerenone on filtration fraction compared to placebo | at baseline and after 3 months on finerenone
  impact of finerenone on filtration fraction compared to placebo
impact of finerenone on total renal vascular resistance compared to placebo | at baseline and after 3 months on finerenone
  impact of finerenone on total renal vascular resistance compared to placebo
impact of finerenone on intraglomerular resistances (resistance of the afferent and efferent arterioles) and intraglomerular pressure (GOMEZ formulae) compared to placebo | at baseline and after 3 months on finerenone
  impact of finerenone on intraglomerular resistances (resistance of the afferent and efferent arterioles) and intraglomerular pressure (GOMEZ formulae) compared to placebo
impact of finerenone on the magnitude of stimulation of renal nitric oxide activity due 318 to L-arginine infusion compared to placebo | at baseline and after 3 months on finerenone
  impact of finerenone on the magnitude of stimulation of renal nitric oxide activity due 318 to L-arginine infusion compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kannenkeril, MD, Principal Investigator — University Hospital Erlangen; Roland E. Schmieder, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- Clinical Research Center Erlangen, Department of Nephrology and Hypertension, University Hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No